CLINICAL TRIAL: NCT03415321
Title: Development of Postnatal Mobile Support Application and Evaluation of the Effectiveness of Mothers' Anxiety and Postpartum Depression Symptoms: Pre-Test Post-Test Randomized Controlled Study
Brief Title: Development of Postnatal Mobile Support Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Vesile KOÇAK, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NecmettinEU
Record Dates: First submitted 2018-01-08; First posted 2018-01-30 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Postpartum Depression; Postnatal Complication; Nurse's Role
Keywords: Postpartum, Nurse, Mothers, Anxiety, Depression, Mobile Support
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with a two-group pre-test and post-test design.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Postpartum Mobile Support Application
  Interventions: Device: Postpartum Mobile Support Application
- Control Group (No Intervention): Routine care

INTERVENTIONS:
Device: Postpartum Mobile Support Application — Women in the experimental group will use the Postpartum Mobile Support Application during six weeks after birth.
  Women will be evaluated three times in total, one for the first day after birth, second for the seventh day after birth and the last for the sixth week after birth.
  Short messages and calls will be remind of women's Postpartum Mobile Support Application use
  Arms: Intervention group

SUMMARY:
A mobile support application will be developed that will support mothers in the postpartum period and will be tested the effects of application on anxiety and depression symptoms.The study will consist of two phases. The first phase of the action research (participant design method) method will be done to provide postpartum mobile support application. In the second stage, postpartum mobile support application will be evaluated for the anxiety and depression symptoms of the mothers after six weeks of use.

DETAILED DESCRIPTION:
The postpartum period is a critical period as it is a unique milestone for many of the important physical, emotional and social changes for parents and newborns (Nilsson, Danbjorg, Larsen, Clemensen, & Kronborg, 2015). In this period, the mother can have problems such as bleeding, infection, pain, breast problems and fatigue. In addition, adaptation to the parenting role, eventual difficulties in adaptating this role and efforts to care for the newborn can reduce the quality of life (WHO, 2012). At the beginning of the postpartum period, mothers need education and support in many subjects such as parenting, baby care, breastfeeding and relevant information and effective care (Ellberg, Hogberg, & Lindh, 2010). The World Health Organization (WHO) also emphasizes the need in the postpartum period suggesting that breastfeeding should be supported, nutrition provided, baby development monitored and family care needs met (WHO, 2013; WHO, 1998).

In recent years, research has shown that postpartum women use information and communication technologies more and more frequently (Gibson & Hanson, 2013) to seek health information (Walker, Im, & Vaughan, 2012). It has been shown that tele-applications for supporting and directing parents in the postnatal period are useful in the transition to parenting in studies from Sweden and Denmark (Lindberg, Christensson, & Öhrling, 2009; Danbjorg, Wagner, & Clemensen, 2014b). Mobile applications providing information on pregnancy health during the prenatal period are widely used (Kennelly, Ainscough, Lindsay, Gibney, McCarthy, & McAuliffe, 2016). It has been shown that it may be possible to meet the support needs of parents by applying innovative communication methods such as online communication at an evidence-based knowledge base. Parents saw the phone application as an informative and navigational lifestyle. Meeting new parents' information needs with chats, knowledge based and automatic messages makes them feel safe and increases their self-sufficiency (Danbjorg, Wagner, & Clemensen, 2014a; Danbjorg, Wagner, & Clemensen, 2014b; Danbjorg, Wagner, Kristensen, & Clemensen , 2015). It is not possible for nurses to be at their mother's side anytime during the whole postpartum period. It is not possible to give all the necessary information without leaving the hospital and transfer the information to practice on the mother's side.

In postpartum period, care needs are increasing so that parents can adapt to their new roles and give effective care to the newborn. It is very important for the mothers to manage this period effectively for their future well-being and relations (Nilsson et. al. 2015). Studies show that mothers and fathers do not get enough postnatal care, do not feel confident with the information they have and feel insecure about what they will do.It is important for parents to feel secure in the postpartum period which in turn will have postive effects on the baby´s health and wellbeing (Danbjorg, Wagner, Kristensen, & Clemensen, 2015; Persson, Fridlund, Kvist, & Dykes, 2011).

Security is defined to feel safe, to be ready, to be satisfied, to feel good and to be sure (Löf et al. 2006, Forster et al 2008, Lindberg et al 2009). Insecurity is a predominant emotion for parents and is characterized by unpredictablity, uncertainity, stress, anxiety, fear, suspicion, feelings of loneliness and despair (George 2005, Forster et al 2008, Hjalmhult and Lomborg 2012). Insecurity is associated with lack of knowledge and skills experienced by parents in newborn care (George 2005, Forster et al 2008, McLachlan et al. 2009). Parents that feel they can manage the baby wellness have sense of security (Löf et al. 2006). They feel safe when they know about the needs of their newborn and aware that they, the parents, are in control of their newborns health (Persson & Dykes 2002). Parents sense of security was associated with the strengthening behaviors they received from health professionals; unity within the family - closeness; autonomy; the mother's physical well-being and the involvement of the father during the birth and the postpartum period (Persson & Dykes, 2002; Persson, Fridlund, & Dykes, 2007; Persson & Dykes, 2009; Persson, Fridlund, Kvist, & Dykes, 2011; Persson, Fridlund, Kvist, & Dykes, 2012).

The postpartum period is a transitional period in which mixed emotions dominate the whole family. In this period, physical symptoms, sleep deprivation, changing demands in work and home life are usually stressful and wearing. Additionally stress anxiety symptomatology has a positive relationship in susceptible people (Moran, Polanin, & Wenzel, 2014). Anxiety usually manifests itself as extreme and persistent fear, anxiety, tension and regularly includes physical symptoms such as sleeping difficulties and lack of focus (Dennis, Falah-Hassani, Brown, & Vigod, 2016). In studies, the anxiety prevalence rates of mothers during the first postpartum year vary between 2% and 45% (Enatescu, et al., 2014; Martini, et al., 2013). Unfortunately, there is increasing evidence that postpartum anxiety affects maternal and infant health negatively. Fatigue, loss of self-esteem and bad body sensations were seen in women who had postpartum anxiety. A deterioration in mother-infant interaction and in sleep patterns, excessive crying and also a deterioration in social relationships was shown. As anxiety acts as a trigger for development of depression, depression is often accompanied by anxiety symptoms (Dennis, Falah-Hassani, Brown, & Vigod, 2016). Depression is a common mental disorder characterized by depressed mood, loss of interest and enjoyment, reduced energy, guilt, low self-esteem, sleep disturbances, decreased appetite and problems in focusing. Depression is a very important health problem for all ages and genders around the world.The World Health Organization (WHO) states that by 2020, depression will contribute to 5.7% of the total illness burden. Depression is the most common type of disease in women (WHO, 2010). For many women, postpartum depression (PPD) usually occurs within the first 12 weeks after birth (Dennis & Dowswell, 2013). PPD is characterized by symptoms consistent with major depressive disorders, bipolar disorders or brief psychotic disorders occurring within 4 weeks of birth (American Psychiatric Association 2013). The symptoms associated with PPD are hopelessness, worthlessness, feelings of guilt, dissatisfaction with one's activities, difficulty in sleeping and concentration and decision-making problems (Gross & Marcussen, 2017). Depressive symptoms in the early postpartum period vary between 5% to 20% in mothers (Patel, Baiely, Jabeen, Ali, Barker, & Osiezagha, 2012; Kerstis, Berglund, Engström, Edlund, Sylven, & Aarts, 2014; O'Hara & McCabe). Dissatisfaction with marriage, antenatal life events, past depressive symptoms, late antenatal depressive symptoms, lack of social support, stressful life events and marital conflicts were identified as potential risk factors for PPD (Dennis, Brown & Morrell, 2016). PPDnegatively affects women's quality of life, close relationships, maternal-infant interactions and infantile and school-age child development outcomes. Early diagnosis and intervention is essential to ensure optimal care for mothers, children and families when short and long term sequels of PPD are considered (McDonald, et al., 2012).

Reducing feelings of loneliness and being lonely, preventing incompatible health behaviors or reactions, increasing individual motivation, providing access to medical services or providing information about benefits, directly affects the development of PPD by supporting health and well-being positively. It is also an indirect means of prevention to identify and reduce the stress factors, increase the number of coping strategies, teaching problem-solving techniques and supporting self-sufficiency (Dennis & Dowswell, 2013). It is clear that there must be a very good support system for all of this to be accomplished. Postpartum support for the mother is of utmost importance (Danbjorg, Wagner, Kristensen, & Clemensen, 2015). "Current social support", including family, friends and health professionals, is one of the factors that mediate the maternal roll (Barclay, Everitt, Rogan, & Schmied 1997; Danbjorg, Wagner, Kristensen, & Clemensen, 2015). In theese studies, it is seen that the support systems of the mothers discharged from hospital after birth are not enough and there is no follow up. The mothers also found it difficult to access the information they need immediately (instantly). Parents were disturbed by the thought that they would disturb nurses when they were looking for help (Danbjorg, Wagner, & Clemensen, 2014a; Danbjorg, Wagner, & Clemensen, 2014b; Danbjorg, Wagner, Kristensen, & Clemensen, 2015). Mothers who are postpartum, spend a lot of time caring for their newborn, but they do not have enough time to get the information they need (Guerra-Reyes, Christie, Prabhakar, Harris, & Siek, 2016). New ways of communicating between healthcare personnel and parents are necessary. More individual timely information increases the self-confidence of mothers (Danbjorg, Wagner, & Clemensen, 2014a; Danbjorg, Wagner, & Clemensen, 2014b; Danbjorg, Wagner, Kristensen, & Clemensen, 2015). In the postpartum period, adequate care and support have been reported to be associated with positive health behaviors and health outcomes, maternal stress reduction and baby health improvement (Guerra-Reyes, Christie, Prabhakar, Harris, & Siek, 2016). There has been no study evaluating the effects of mobile support application on postpartum sense of security, anxiety and depression during the postpartum period.

Conceptual framework of the study Orem's Self-care Deficit Nursing Theory is used as the conceptual framework of this study. Acording to Orem people have a natural ability for self care and that nursing should focus on affecting that ability there is a constant need for strength and energy in order for a person to move on with his life and ability. The person has the power to self-care for her/himself and others and to determine their needs. The self-care skill required to maintain the life and function of the adult person varies from person to person. The person explores and develops different ways in describing the requirements for himself and others, and the necessary power in total. People who live together and share their responsibilities as a group are held accountable for the care of both themselves and others suffering from inadequate self-care (Orem, 2001, Fitzpatrick & Whall, 1996). The self-care of mothers who do not receive accurate health information may be affected. Likewise, the health of the children of mothers who do not get enough information is affected.

ELIGIBILITY:
Inclusion Criteria:

* Giving birth full term 39 weeks 0 days and 40 weeks 6 days (ACOG 2013)
* Having a phone with Android feature and having an internet connection
* Baby's normal birth weight and having APGAR score 8 and above

Exclusion Criteria:

* Adolescent pregnants
* Having anxiety and depression
* Complication developments in the mother or newborn after delivery
* Newborn stay in the intensive care unit
* Visually impaired, hearing impaired

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 124 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | Postpartum 6 weeks
  Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report scale that evaluates depressive symptoms just after delivery developed by Cox et al. (1987). EPDS will be used to assess depression in fathers and mothers. Each item is scored on a four-point scale(0-3), the minimum and maximum scores being 0 and 30,respectively. The prevalence of depression will be identified using the recommended cut-off point of 13 or above. The following severity ranges were established for the EPDS: None or minimal depression (0-6), Mild depression (7-13), Moderate depression (14-19), Severe depression (19-30).The EPDS score should not override clinical judgment. A careful clinical assessment should be carried out to confirm the diagnosis.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory | Postpartum 1th day and 6 weeks
  State-Trait Anxiety Inventory (STAI) is self-report questionnaire consists of two subscales each containing 40 items, 20 items allocated to each of the S-Anxiety and T-Anxiety subscales. It has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale. Higher scores indicate greater anxiety. The scores obtained from the scale range theoretically from 20 to 80. Bigger score indicates high anxiety level; small score indicates low anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Vesile KOÇAK, Principal Investigator — Researcher
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Kocak V, Ege E, Iyisoy MS. The development of the postpartum mobile support application and the effect of the application on mothers' anxiety and depression symptoms. Arch Psychiatr Nurs. 2021 Oct;35(5):441-449. doi: 10.1016/j.apnu.2021.06.009. Epub 2021 Jun 22. PMID 34561057